CLINICAL TRIAL: NCT04948580
Title: Reducing Violence by Teachers Against Children: A Multi-Site Cluster Randomized Controlled Trial of Interaction Competencies With Children - for Teachers (ICC-T) in Primary and Secondary Schools in Tanzania, Uganda and Ghana
Brief Title: Preventing Violence by Teachers Against Children in Sub-Saharan Africa
Acronym: EVIDENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bielefeld University (Other)
Collaborators: Daressalaam University College of Education (DUCE) (Unknown); Mbarara University of Science and Technology (MUST) (Unknown); Presbyterian University College Ghana (PUCG) (Unknown)
Responsible Party: Principal Investigator, Tobias Hecker, PhD, Principal Investigator, Bielefeld University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HE 8505/1-1
Record Dates: First submitted 2021-06-28; First posted 2021-07-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Violence by Teachers
Keywords: school violence; teacher violence; intervention; teachers; students; primary schools; secondary schools

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICC-T (Experimental): 5.5 days with 8 hours of training for teachers aiming at changing attitudes towards violence and equipping teachers with non-violent discipline strategies
  Interventions: Behavioral: Interaction Competencies with Children - for Teachers (ICC-T)
- Monitoring condition (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Interaction Competencies with Children - for Teachers (ICC-T) — Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting
  Arms: ICC-T

SUMMARY:
Violence has severe and long-lasting negative consequences for children's and adolescents' well-being and psychosocial functioning, thereby also hampering communities' and societies' economic growth. Studies show high prevalence of violence by teachers against children in Sub-Saharan Africa, both in countries where violence is lawful as disciplinary measure at school and in countries where it has been officially banned. In addition to legal and structural factors (e. g. stressful working conditions for teachers), attitudes favoring violence against children as an effective and acceptable discipline method and the lack of access to alternative non-violent strategies are likely to contribute to teachers' ongoing use of violence against children.

Notwithstanding, there are currently very few school-level interventions to reduce violence by teachers that a) have been scientifically evaluated and b) that focus both on changing attitudes towards violence and on equipping teachers with non-violent discipline strategies.

Thus, the present study tests the effectiveness of the preventative intervention Interaction Competencies with Children - for Teachers (ICC-T) in primary and secondary schools in Tanzania, Uganda and Ghana. Previous studies have provided initial evidence on the feasibility and effectiveness of ICC-T to reduce teacher violence in primary and secondary schools in Tanzania and secondary schools in Uganda. This study aims to provide further evidence for the effectiveness of ICC-T to reduce violence and to improve children's functioning (i.e. mental health, well-being, academic performance) across educational settings, societies and cultures.

DETAILED DESCRIPTION:
The study is a multi-site cluster randomized controlled trial with schools (clusters) as level of randomization. Multi-stage random sampling will be applied to select three zones per country (Tanzania, Uganda and Ghana) and one district in each zone. In each district, eight public schools will be randomly selected, resulting in a total number of 72 schools (24 per country). Schools will be stratified based on school type (primary or secondary school) and location (rural or urban), leading to 36 sites or cluster pairs (3 countries x 3 zones x 2 school types x 2 locations). In each site, one school will be randomly allocated to the intervention group (that will receive the ICC-T intervention) and one school to the control group (that will receive no intervention).

At each school, 40 students (stratified by gender) in the third year of primary school or in the first year of secondary/junior high school and all teachers (expected average number: 20) will be recruited. Thus the final sample will comprise 2880 students and at least 1440 teachers.

The study will have three data assessment points: baseline assessment prior to the intervention, the first follow-up assessment six months after the intervention and the second follow-up assessment 18 months after the intervention. In addition, feasibility data will be assessed in the intervention group at the beginning and the end of the intervention.

Primary outcome measures are student- and teacher-reported physical and emotional violence by teachers in the past week. Secondary outcome measures include teachers' attitudes towards violence against students, children's emotional and behavioral problems, quality of life, and cognitive functioning.

ELIGIBILITY:
General:

Inclusion Criteria:

* All: Written informed consent (if underaged by parents (written) & minors themselves (oral or written)
* Students: Enrollment in class 3 of primary school or in class 1 of secondary school
* Teachers: All teachers employed at the school

Schools:

* Public schools
* Mixed-gender schools
* Day schools
* At least 40 students in selected class/stream

Exclusion criteria:

* Acute drug or alcohol intoxication
* Acute psychotic disorder

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3264 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change of students' exposure to emotional and physical violence by teachers | The CTS will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention).
  The Conflict Tactics Scale (CTS) will be used to assess students' self-reported experiences of emotional and physical violence by teachers at school in the past week. Higher scores indicate higher levels of violence that is used by teachers. A change of exposure to violence in the intervention group is hypothesized.
Change of teachers' use of emotional and physical violence | The CTS will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention)
  The Conflict Tactics Scale (CTS) will be used to assess teachers' use of emotional and physical violent discipline measures against students in the past week. Higher scores indicate higher levels of violence that is used by teachers. A change in the use of violence in the intervention group is hypothesized.

SECONDARY OUTCOMES:
Change of teachers' positive attitudes towards emotional and physical violence | The adapted version of CTS will be used at T 1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after the intervention).)
  Teacher's attitudes towards emotional and physical violence will be assessed with an adapted version of the Conflict Tactic Scale (CTS). Higher scores indicate higher levels of positive attitudes towards violence. A change of positive attitudes towards violence in the intervention group is hypothesized.
Change of student's mental health | The PSC-Y will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention)
  The Pediatric Symptom Checklist - Youth Report (PSC-Y) will assess students' emotional and behavioral problems. Higher scores indicate higher levels of students' mental health problems. A change of mental health problems in the intervention group hypothesized.
Change of students' quality of life | The KIDSCREEN-10 will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention) ]
  The KIDSCREEN-10 will assess students' quality of life. Higher scores indicate higher levels of students' quality of life. A change of quality of life in the intervention group is hypothesized.
Change of students' cognitive functioning | The Psych Lab 101 application will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention)
  Four tasks implemented in the Android application Psych Lab 101 (Neurobehavioral Systems, 2020) will be used to assess children's cognitive abilities including selective attention, working memory, interference control and cognitive control. Higher scores indicate higher levels of students' cognitive abilities. A stronger improvement of cognitive functioning in the intervention group compared to the control group is hypothesized.

OTHER OUTCOMES:
Change of students' academic performance | The standardized achievement tests will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention).
  Purpose-built tests will be used to assess students' numeracy and literacy skills. Higher scores indicate higher levels of students' academic skills. In addition, students' grades in the previous term's exams will be obtained from the school administration. A change in academic performance in the intervention group is hypothesized.
Change of students' social competence | The Social Cognitive Map Technique - peer nomination will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention).
  The Social Cognitive Map Technique will assess students' social competence through peer nominations. Higher scores indicate higher levels of students' social competence. A change of social competence in the intervention group is hypothesized.
Change of peer victimization | The MPVS-24 will be used at T1 (baseline, prior to intervention), T2 (first follow-up, 6 months after intervention) and T3 (second follow-up, 18 months after intervention).
  The Multidimensional Peer Victimization Scale (MPVS-24; Joseph & Stockton, 2018) assesses children's experiences of violence by peers using the 24-item version. A change of exposure to violence in the intervention group is hypothesized.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hecker, Prof. Dr., Principal Investigator — Bielefeld University
Locations (3):
- Presbyterian University College Ghana, Abetifi, Ghana
- Daressalaam University College of Education, Dar es Salaam, Tanzania
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scharpf F, Kirika A, Masath FB, Mkinga G, Ssenyonga J, Nyarko-Tetteh E, Nkuba M, Karikari AK, Hecker T. Reducing physical and emotional violence by teachers using the intervention Interaction Competencies with Children - for Teachers (ICC-T): study protocol of a multi-country cluster randomized controlled trial in Ghana, Tanzania, and Uganda. BMC Public Health. 2021 Oct 24;21(1):1930. doi: 10.1186/s12889-021-11950-y. PMID 34689732